CLINICAL TRIAL: NCT03391687
Title: Investigation of Incidence of Pancreatic Fistula After Radical Gastrectomy in Gastric Cancer Patients
Brief Title: Incidence of Pancreatic Fistula After Radical Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSGC-003
Record Dates: First submitted 2017-12-15; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer; Pancreatic Fistula; Complication
Keywords: Gastric Cancer; Pancreatic Fistula; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amylase Test: gastric cancer patients receiving radical gastrectomy
  Interventions: Diagnostic Test: Amylase Test

INTERVENTIONS:
Diagnostic Test: Amylase Test — body fluid amylase will be tested after radical gastrectomy in scheduled interval

SUMMARY:
This study is designed to investigate the incidence of pancreatic fistula after radical gastrectomy in gastric cancer patients.

DETAILED DESCRIPTION:
Pancreatic fistula, which can lead to fatal end, is one of the most serious complications after radical gastrectomy. It is usually treated as a key factor to evaluate the quality of gastrectomy. The incidence of pancreatic fistula is far different between different areas, knowing the prevalence of pancreatic fistula and risk factors can help us to prevent pancreatic fistula and improve the short time outcome of gastric cancer surgery treatment. So, we designed this perspective, multi-center study to investigate the incidence of pancreatic fistula and its outcome in China.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed stomach adenocarcinoma
* preoperative curatively resectable tumor

Exclusion Criteria:

* pancreas resection
* emergent surgery due to gastric cancer acute complications
* cancer of gastric remnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: stomach adenocarcinoma patients who recieved radical gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pancreatic Fistula | in 30 days following gastrectomy
  the incidence of pancreatic fistula after radical gastrectomy in gastric cancer patients

SECONDARY OUTCOMES:
The Classification of Pancreatic Fistula | in 30 days following gastrectomy
  the percentage of different grades of pancreatic fistula, including Grade BL, Grade B and Grade C
The mortality of Grade B and C Pancreatic Fistula | in 30 days following gastrectomy
  the percentage of patients died of Grade B or C pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Fenglin Liu, MD, Principal Investigator — Fudan University
Locations (20):
- China (20):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - South West Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Weifang People's Hospital, Weifang, Shandong
  - ZhongShan hospital Fudan university, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ruijing Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicince, Hangzhou, Zhejiang

REFERENCES:
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Yu HW, Jung DH, Son SY, Lee CM, Lee JH, Ahn SH, Park DJ, Kim HH. Risk factors of postoperative pancreatic fistula in curative gastric cancer surgery. J Gastric Cancer. 2013 Sep;13(3):179-84. doi: 10.5230/jgc.2013.13.3.179. Epub 2013 Sep 30. PMID 24156038
- [Background] Tanaka K, Miyashiro I, Yano M, Kishi K, Motoori M, Seki Y, Noura S, Ohue M, Yamada T, Ohigashi H, Ishikawa O. Accumulation of excess visceral fat is a risk factor for pancreatic fistula formation after total gastrectomy. Ann Surg Oncol. 2009 Jun;16(6):1520-5. doi: 10.1245/s10434-009-0391-y. Epub 2009 Mar 8. PMID 19267237
- [Background] Jiang X, Hiki N, Nunobe S, Kumagai K, Nohara K, Sano T, Yamaguchi T. Postoperative pancreatic fistula and the risk factors of laparoscopy-assisted distal gastrectomy for early gastric cancer. Ann Surg Oncol. 2012 Jan;19(1):115-21. doi: 10.1245/s10434-011-1893-y. Epub 2011 Jul 8. PMID 21739317
- [Background] Kobayashi D, Iwata N, Tanaka C, Kanda M, Yamada S, Nakayama G, Fujii T, Koike M, Fujiwara M, Kodera Y. Factors related to occurrence and aggravation of pancreatic fistula after radical gastrectomy for gastric cancer. J Surg Oncol. 2015 Sep;112(4):381-6. doi: 10.1002/jso.24001. Epub 2015 Aug 8. PMID 26256914
- [Background] Komatsu S, Ichikawa D, Kashimoto K, Kubota T, Okamoto K, Konishi H, Shiozaki A, Fujiwara H, Otsuji E. Risk factors to predict severe postoperative pancreatic fistula following gastrectomy for gastric cancer. World J Gastroenterol. 2013 Dec 14;19(46):8696-702. doi: 10.3748/wjg.v19.i46.8696. PMID 24379588
- [Background] Kung CH, Lindblad M, Nilsson M, Rouvelas I, Kumagai K, Lundell L, Tsai JA. Postoperative pancreatic fistula formation according to ISGPF criteria after D2 gastrectomy in Western patients. Gastric Cancer. 2014;17(3):571-7. doi: 10.1007/s10120-013-0307-1. Epub 2013 Oct 9. PMID 24105422
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309